CLINICAL TRIAL: NCT06035900
Title: Phase 1, Open-Label, One-Treatment, Single-Dose, One-Period, Pharmacokinetic Study of Psilocin 4 mg as Its Mucic Acid Salt (L-130) Form, in Healthy Subjects Under Fasted Conditions
Brief Title: Evaluation of Safety, Rate and Extent of Absorption of Psilocin Mucate
Acronym: Psilocin-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lobe Sciences Ltd. (Industry)
Collaborators: Pharmaceutical Research Unit, Jordan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PSIL22060
Record Dates: First submitted 2023-08-31; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Side Effect of Drug
MeSH Terms: interventions — psilocin

STUDY DESIGN:
Intervention Model Description: The aim of the study is to assess the bioavailability and pharmacokinetic parameters and to monitor the safety and tolerability of a formulation in healthy subjects under fasting conditions after a single oral dose of L-130 Capsules containing 2 mg of psilocin as its Mucic Acid Salt or Conjugate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10 normal healthy male volunteers (Experimental): 10 normal healthy male volunteers where each subject was given an identification code after signing the informed consent which was obtained according to APIC/PRU procedure of obtaining Consent form. The identification code consisted of the subject's initials, and a serial number.
  Interventions: Drug: Psilocin

INTERVENTIONS:
Drug: Psilocin — single 4mg dose of psilocin mucate was administered to healthy 10 volunteers
  Other Names: Psilocin Mucate

SUMMARY:
Psilocin is the active metabolite of psilocybin a natural material found in several types of fungi. The bioavailability of psilocybin, the prodrug of psilocin, has been reported to be over 60%. However, pharmacokinetics and bioavailability of psilocin mucate has not been reported. This Phase I "First in Man" study of psilocin mucate is designed to determine its safety, pharmacokinetics, and bioavailability. The study is conducted under the supervision of physicians and psychiatrists who also will administer a mini-mental state evaluation and report observable anti-anxiolytic effect of the dosage. Safety and possible indications of efficacy will be tracked during the study period, a week following the dose administration and one month after.

DETAILED DESCRIPTION:
This study is designed to assess the bioavailability and pharmacokinetic parameters and to monitor the safety and tolerability of Psilocin 2 mg as its Mucic Acid Salt (L-130) form, a proprietary drug candidate of Lobe Sciences Ltd., in healthy subjects under fasted conditions.

The study will be conducted in compliance with the protocol and applicable regulatory requirements, GCP and GLP principles and guidelines: Declaration of Helsinki as amended by the 64th WMA General Assembly, Fortaleza, Brazil, November 2013, FDA Guidelines for Bioavailability & Bioequivalence Studies and OECD Principles of Good Laboratory Practice will be observed.

The study population will consist of 10 Healthy Subjects aged between 21 and 50 years (inclusive), body mass index 18.5 to 30.0 kg/m2 inclusive (minimum of 50 kg weight for males and 45 kg for females), nonsmokers or quit smoking 24 hours prior to dosing.

The investigational test product L-130 Capsules containing 2 mg of psilocin as its Mucic Acid Salt of Lobe Sciences Ltd. consisted of single oral dose containing 2 mg of Psilocin (equivalent to 4 mg as Psilocin Mucate salt).

Each dose will be administered orally, with 240 mL of water in sitting position under sodium light to healthy subjects after an overnight fast of at least 10 hours in the morning of study dosing day. The study will be conducted as an open label study. Therefore, blinding will not be done. However, the bioanalysis will be performed blinded with regard to the sequence of product administration. Each subject will have a pre-dose sample of 8 ml collected and 13 additional 8 ml samples collected over a 24 hour period.

The principal and/ or clinical investigator and study staff will monitor subjects throughout the hospitalization periods. Blood pressure and heart rate will be measured before dosing and at scheduled intervals after dosing. The principal and/ or clinical Investigator will be available throughout each hospitalization period. During outpatient phases, study staff will be available during regular working hours.

Subjects' safety will be observed at scheduled intervals of before dosing (-1.00) and 0.50, 0.75, 1.00, 2.00, 3.00, 5.00, 8.00, 12.00, 16.00 and 24.00 hours after drug administration. Subjects will be queried on adverse events. In addition, voluntary reporting of adverse events by subjects will be reported.

Mini Mental State Examination (MMSE) score will be assessed to dosed subjects by CI/PI approximately two hours after drug administration, and the results will be tabulated in the final report. Subjects will be asked to report changes in their mood, or other observations during and following the study period. Subjects will also be followed up by phone call after one week and four weeks of dosing to assess if they are experiencing changes in feeling or having improved mood, and the outcomes of the phone calls will be tabulated in the final report.

Following the collection of blood samples and appropriate processing, each sample will be analyzed with a validated analytical method to determine the pharmacokinetic profile of psilocin mucate in plasma.

All clinical laboratories test results of screening lab tests will be summarized by descriptive statistics. Follow up lab tests will also be summarized by descriptive statistics.

The aim of the study is to assess the bioavailability and pharmacokinetic parameters and to monitor the safety and tolerability of the formulation in healthy subjects under fasting conditions after a single oral dose of L-130 Capsules containing 2 mg of psilocin as its Mucic Acid Salt. The final report will provide safety, tolerability and pharmacokinetics of the test product. The study will also report patient reported pharmacology.

ELIGIBILITY:
Inclusion Criteria:

Age 21-50 years. Body-mass index 18.5 to 30.0 kg/m2 inclusive. (Minimum of 50 kg weight for males and 45 kg for females).

Subject is available for the whole study period and gave written informed consent.

Normal physical examination or being assessed as clinically non-significant by the attending physician.

Normal neurological, cardiovascular, cerebrovascular, gastrointestinal and respiratory systems.

Normal Vital Signs. Normal Electrocardiogram (ECG). Subjects refraining from alcohol use, other study medication and drugs.

Lab test inclusion criteria:

On Screening Chemistry, Hematology and Urine laboratory screening results within the normal range, or being assessed as clinically non-significant by the attending physician.

Normal Liver and kidney function test.

Exclusion Criteria:

Lab test exclusion criteria

On screening

1. Positive serology test.
2. Chemistry, Haematology and Urine laboratory screening results not within the normal range, or being assessed as clinically significant by the attending physician
3. Abnormal Liver and kidney function test.
4. Positive hCG for female subjects.

On Admission:

1. The intake of caffeine, xanthene, or CO2-containing beverages within 24 hours of drug administration.
2. Consumption of alcohol, grapefruit or grapefruit containing products within 7 days of drug administration
3. Ingestion of any supplements like vitamins or herbal products within 7 days prior to each drug administration study.
4. Clinically significant illness 4 weeks before study Period I
5. Exhausting physical exercise in the last 24 hours (e.g. weight lifting) or any recent significant change in dietary or exercise habits.
6. Abnormal vital signs and being assessed as clinically significant.
7. Vomiting, diarrhea on admission.
8. Subjects with concurrent medication must be taken 14 days before drug administration and during study period especially warfarin, aspirin, non-steroidal anti-inflammatory drugs, levodopa, antipsychotic medicinal products, fibrates, ciclosporin, fusidic acid (a medicine for bacterial infection), orally and or by injection.
9. Participation in another bioequivalence study and/or clinical trials within 80 days prior to the start of this study Period.
10. Have been taking medication that could affect the investigated drug product: a) Regular consumption of drugs during the b) consumption of enzyme stimulating or inhibiting drugs (e.g.

    Barbiturates, Carbamazepine, Phenytoin, Amphetamine, Benzodiazepine, cannabinoid, cocaine, opiates, phencyclidine and methadone) during two weeks before the study initiation.
11. Subject taking medications that belongs to strong CYP3A4 inhibitors (including, but not limited to, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir) or inducers (e.g., phenytoin, rifampicin, carbamazepine, phenobarbital and St. John's Wort) within 4 weeks prior to study.
12. Subject taking monoamine oxidase inhibitors medications.
13. Subject taking selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitors (SSRI/SNRI) medications.
14. Subject taking uridine diphosphate glucuronosyl transferase enzyme modulators medication.

Pre-dose:

1. Pre-dosing blood pressure less than 110/70 mmHg.
2. Pre-dosing heart rate less than 70 beats per minute.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Determination of adverse events | 28 days
  Frequency

OTHER OUTCOMES:
Plasma Concentration (Cmax) | 24 hours
  nanograms/milliliter (ng/ml)
Area Under the plasma concentration versus time curve (AUC) | 24 hours
  nanograms minute/milliliter (ng min/ml)
Time to maximum plasma concentration (Tmax) | 24 hours
  minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Abdulkhaleq, MD, Principal Investigator — Arab Pharmaceutical Industry Pharmaceutical Research
Locations (1):
- Pharmaceutical Research Unit, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the bioavailability data and pharmacokinetics of psilocin mucate in a peer reviewed publication. We also plan to share safety information gathered during the Phase 1 segment of the trial also in a separate publication in a peer reviewed journal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: We hope to complete the trial and receive a final report that will be the source of at least two publications in or around March 2024.
Access Criteria: We plan to share the data from the pharmacokinetics study with any academic research or medical institution upon written request to the Project Leader and Central Contact Person: Dr. Fred D. Sancilio